CLINICAL TRIAL: NCT04120311
Title: Phase I Study of Sequestered Transscleral, Controlled-Release Dexamethasone Delivered Via Episcleral Reservoir for Treatment of Macular Edema & Inflammatory Disorders of the Eye Posterior Pole Including Sclera, Choroid, Retina or Vitreous
Brief Title: Episcleral Dexamethasone for Treatment of Macular Edema and Inflammatory Disorders of the Posterior Pole
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Targeted Therapy Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3TDEX-02
Record Dates: First submitted 2019-10-03; First posted 2019-10-09 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Macular Edema; Radiation Retinopathy; Branch Retinal Vein Occlusion; Epiretinal Membrane; Central Serous Retinopathy With Pit of Optic Disc; Commotio Retinae; Vitritis
Keywords: Macular Edema; Radiation Retinopathy; Branch Retinal Vein Occlusion; Epiretinal Membrane; Central Serous Retinopathy with Pit of Optic Disc; Commotio Retinae; Vitritis
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion; Epiretinal Membrane; Uveitis, Intermediate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase I open label study (Experimental): Drug: Episcleral Dexamethasone Sequestered Transscleral, Controlled-Release Dexamethasone
  Other Names:
  • Sustained Release Transscleral Dexamethasone
  Interventions: Drug: Episcleral Dexamethasone

INTERVENTIONS:
Drug: Episcleral Dexamethasone — Sustained Release Episcleral Dexamethasone
  Other Names: Sequestered Transscleral, Controlled-Release Dexamethasone; Sustained Release Transscleral Dexamethasone

SUMMARY:
This phase I trial will assess primarily the safety and secondarily anti-inflammatory effect of Episcleral Dexamethasone in patients suffering from macular edema and other disorders of the retina, choroid and vitreous.

DETAILED DESCRIPTION:
This phase I trial will assess primarily the safety and secondarily anti-inflammatory effect of Episcleral Dexamethasone in patients suffering from macular edema and other disorders of the retina, choroid and vitreous. Numerous studies have documented the anti-inflammatory activity of Dexamethasone in macular edema associated with diabetes, branch retinal vein occlusion, and non-infectious posterior uveitis. The investigators hypothesize that Episcleral Dexamethasone is safe, tolerable and that its anti-inflammatory activity will interface with the pro-inflammatory cascade associated with macular edema due to diabetes, surgery, trauma, vein occlusions, uveitis and retinal degeneration to improve visual structure and function. The investigators hypothesize that Episcleral Dexamethasone is safe, tolerable and that its anti-inflammatory activity will reduce macular edema and improve vision. The investigator's objective is to primarily assess the safety, tolerability and pharmacokinetics of Episcleral Dexamethasone in patients with macular edema; to secondarily assess efficacy in reducing macular edema and improving visual structure and function. The main outcome of the study is safety assessment. Secondary outcomes are assessment of visual acuity and anatomical changes in the macula as measured via optical coherence tomography (OCT) and fluorescein angiogram.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years;
* Visual acuity letter score in study eye < 70 and ≥ 25 letters (approximate Snellen equivalent 20/32 to 20/320);
* Ophthalmoscopic evidence of center-involved macular edema, within the central subfield (CSF);
* Inflammatory disorders of the sclera, choroid, retina or vitreous

Exclusion Criteria:

* Inability to understand informed consent, cooperate with testing or return to follow up visits;
* Pregnant or lactating women;
* Co-existent ocular disorder of the cornea, lens or media that will interfere with assessment of safety or efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
A primary outcome measure of the study is ocular safety assessment as measured by comprehensive ophthalmic exam. | 12 Months
  Assessment of ocular safety as measured by comprehensive ophthalmic exam.

SECONDARY OUTCOMES:
A secondary outcome is assessment of visual acuity. | 12 Months
  Secondary outcome is assessment of visual acuity.
A secondary outcome is assessment of anatomical changes in the macula as measured via optical coherence tomography (OCT). | 12 Months
  A secondary outcome is assessment of anatomical changes in the macula as measured via optical coherence tomography (OCT).

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Leng, MD, Principal Investigator — Stanford Medicine
Locations (1):
- Stanford Medicine Ophthalmology, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romano F, Lamanna F, Gabrielle PH, Teo KYC, Battaglia Parodi M, Iacono P, Fraser-Bell S, Cornish EE, Nassisi M, Viola F, Agarwal A, Samanta A, Chhablani J, Staurenghi G, Invernizzi A. Update on Retinal Vein Occlusion. Asia Pac J Ophthalmol (Phila). 2023 Mar-Apr 01;12(2):196-210. doi: 10.1097/APO.0000000000000598. Epub 2023 Feb 14. PMID 36912792